CLINICAL TRIAL: NCT02019433
Title: Post Market Clinical Follow-Up of Acetabular Titan-Augment Structan®
Status: Terminated | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1212
Record Dates: First submitted 2013-12-05; First posted 2013-12-24 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Total Hip Arthroplasty Revision
Keywords: THA, augment, revision, pelvis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Structan®
  Interventions: Device: Structan®

INTERVENTIONS:
Device: Structan®

SUMMARY:
Implant Survival as well as clinical and radiological Follow-Up of acetabular Titan-Augment Structan®

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years
* Indication for cementless hip arthroplasty with acetabular defects that need Allograft or titanium augment
* Patient consent for study participation
* Physical and mental willingness to participate in the follow-ups

Exclusion Criteria:

* Patient not available for follow-up
* Increased anesthetics risks for the patient according to the "American Society of Anesthesiology": ASA IV
* Tumor
* Alcohol- or Drug abuse
* Permanent cortisone therapy
* Clinically relevant infection
* (Planned) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: specialist clinical centre
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Implant Survival Rates | 12 months
  Implant survival is analysed at follow-up examinations at 3 and 12 months

SECONDARY OUTCOMES:
Clinical Outcome | 3 and 12 months
  Harris Hip Score
Pain | 3 and 12 months
  Visual Analogue Scale (VAS)
Osteolysis | 3 and 12 months
  Radiographic Outcome
Ossifications | 3 and 12 months
  Radiographic Outcome
Implant Position | 3 and 12 months
  Radiographic Outcome
Migration of Structan® | 3 and 12 months
  Radiographic Outcome

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Charite Campus Berlin Mitte, Berlin
  - Klinik am Eichert, Göppingen
  - St. Remigius Krankenhaus Opladen, Leverkusen